CLINICAL TRIAL: NCT02069886
Title: A Multicenter, Open-label, Single Arm, Interventional Phase IV Study, to Evaluate the Effect of Deferasirox on Endocrine Complications in Subjects With Transfusion Dependent Thalassemia
Brief Title: Effect of Deferasirox on Endocrine Complications in Subjects With Transfusion Dependent Thalassemia
Acronym: CENTAurus
Status: Withdrawn | Phase: Phase 4 | Type: Interventional
Sponsor: Novartis Pharmaceuticals (Industry)
Responsible Party: Sponsor
Organization: Novartis (Industry)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: CICL670AIT12
Record Dates: First submitted 2014-02-20; First posted 2014-02-24 (Estimated); Last update posted 2017-04-20 (Actual); Status verified 2015-03

CONDITIONS: Thalassemia (Transfusion Delendent)
Keywords: Endocrine complications; transfusion dependent thalassemia
MeSH Terms: conditions — Thalassemia | interventions — Deferasirox

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- deferasirox (Experimental): single arm. all patients will receive deferasirox
  Interventions: Drug: deferasirox

INTERVENTIONS:
Drug: deferasirox — 125, 250, 500 mg dispersable tablets

SUMMARY:
The CENTAurus trial is a prospective clinical study designed to address systematically some of the relevant endocrine complications in an iron overloaded thalassemic population, primary objective being the assessment of the effect of deferasirox therapy on glucose metabolism/homeostasis. Other endocrine parameters complementary or supportive to the primary objective will be assessed and analyzed during this study. A number of lab parameters related to other axes of the endocrine system will be collected and analyzed.

ELIGIBILITY:
Inclusion Criteria:

1. Beta thalassemia major and severe intermedia patients transfusion dependent and with transfusional iron overload 2. Patients with diagnosis of impaired fasting glucose or impaired glucose tolerance 4.Patients naïve to deferasirox or patients who already receive deferasirox at sub-optimal doses 5.Cardiac MRI T2* >10 msec; 7.normal cardiac function (LVEF > 56%);

Exclusion Criteria:

1. Non transfusional hemosiderosis;
2. Patients with diabetes mellitus (genetic or secondary) or history of diabetes mellitus in 1st degree relatives;

4.Patients who received organ transplant; 5.Patients with galactose intolerance, severe lactase deficiency or glucose-galactose malabsorption; 6.Patients unable to tolerate (or who have unacceptable toxicities to) prior treatment with deferasirox; 7.History of hypersensitivity to the study drug or any of its excipients; 8. Renal impairment 10. Liver impairment; 11.Patients with active chronic hepatitis B infection, active hepatitis C infection;

Other protocol-defined inclusion/exclusion criteria may apply" at the end

Ages: 2 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 0 (Actual)
Dates: Start 2014-12; Primary Completion 2018-12 (Estimated); Study Completion 2018-12 (Estimated)

PRIMARY OUTCOMES:
Change from baseline of glucose blood level measured after 2 h after receiving a glucose-equivalent oral challenge | 36 months
  The primary efficacy variable is the change (mg/dl) from baseline to 36 months of glucose plasma levels measured 2 hr post glusose equivalent oral challange.
  After a 12-hour overnight fasting, at zero time (baseline) blood sample will be drawn and afterwards patients will receive a glucose-equivalent oral challenge (75 grams). After glucose loading plasma samples will be drawn at 30, 60, 90, 120 minutes for determination of plasma glucose. This will be repeated every 6 month till end of study

SECONDARY OUTCOMES:
Glucose of OGTT ( AUC) | baseline and every 6 months measurement of 2hour Glocose of OGTT
  change in of glucose metabolism during deferasirox treatment measuring the change versus baseline of 2-hr and fasting glucose plasma level of OGTT.After a 12-hour overnight fasting, at zero time (baseline) blood sample will be drawn and afterwards patients will receive a glucose-equivalent oral challenge (75 grams). After glucose loading plasma samples will be drawn at 30, 60, 90, 120 minutes for determination of plasma glucose . This will be repeated every 6 months till end of study
change on insulin secretion and sensitivity | baseline and every 6 months measurement of 2hr Glucose OGTT
  Change in insulin secretion and insulin sensitivity at every measurement versus screening. Stumvol Formula will be applied to values of 2hr glucose OCTT to calucolate insulin secretion and insulin sensitivity. After a 12-hour overnight fasting, at zero time (baseline) blood sample will be drawn and afterwards patients will receive a glucose-equivalent oral challenge (75 grams). After glucose loading plasma samples will be drawn at 30, 60, 90, 120 minutes for determination of insulin concentration.
Measurement of thyroid hormones TSH and FT4 | baseline and every 12 months
  Changes in plasma levels of TSH and FT4 at every measurement versus screening. Blood samples will be drawn from the patient at baseline and every 12 month till end of study and plansa concentration of thyroid hormons TSH and FT4 will be assessed.
Risk factors for the impairment of glucose homeostasis | baseline and monthly till End of Study
  information on age, sex, ethnicity, BMI, metabolic syndrome (hypertension, dyslipidemia, hypertrygliceridemia), chronic use of steroids, use of immunosuppressive drugs, growth hormonal deficit will be collected on a monthly basis till end of study
Changes in endocrine funcionts parameters | baseline and monthly till EOS
  - Female patients will be assessed for the presence or absence of menses every month versus baseline .Use of current hormonal replacing therapy, if any (e.g. thyroxin therapy for patients with non-compensated hypothyroidism, hormonal replacement drugs for hypogonadal patients) will be checked on a monthly basis versus baseline
Changes in parameters of bone metabolism | baseline, monthly or every 6 months till end of study
  - Blood samples wiil be drawn to measure levels of serum calcium, phosphorus, alkaline phosphatase, vitamin D levels (25-hydroxycholecalciferol), serum calcium, parathormone (intact 1-84 PTH) from baseline to the end of study. Blood samples will be drawn to assess also Vitamin D and parathormone at baseline and then every six months. The intact parathormone will be assessed by evaluating the 1-84 PTH form. Inorganic phosphorus, serum calcium will be assessed at baseline and then monthly; alkaline phosphatase will be evaluated at baseline, every two weeks during the first month of treatment and monthly thereafter till EOS.
Iron overload status | baseline and regularly till end of study (monthly or yearly as specified)
  Blood samples will be drawn to assess Serum Ferriting. Liver and cardiac iron will be assessed by MRI (MRI R2 annual measurements for liver, MRI T2* annual measurements for cardiac); -Relationship between changes in SF, LIC and cardiac T2* and changes in primary (OGTT) and secondary endpoints (glucose metabolism trend, insulin secretion and insulin sensitivity);
Safety of deferasirox therapy | baseline and at every scheduled visit (weekly for the first months or after dose escalation and monthly thereafter or yearly till EOS
  Clinical and laboratory monitoring of AEs and SAEs (in particular changes in hepatic, renal, audiometric and ophthalmology parameters). Blood samples will be drawn to assess liver functions, renal funtions. Urine test will be performed to assess renal functions. An audiometric and ophalmologic visit will be done to assess eyes and ears functions.

CONTACTS AND LOCATIONS:
Overall Officials: Novartis Pharmaceuticals, Study Director — Novartis Pharmaceuticals